CLINICAL TRIAL: NCT03194334
Title: Effect of a 6-month Vegetarian Diet in Omnivorous Women on Body Creatine, Carnitine and Carnosine Stores
Brief Title: Creatine, Carnitine and Carnosine in Vegetarians
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: EC/2012/666
Record Dates: First submitted 2017-06-15; First posted 2017-06-21 (Actual); Results first posted 2019-02-28 (Actual); Last update posted 2019-02-28 (Actual); Status verified 2018-10

CONDITIONS: Dietary Modification
Keywords: vegetarianism; creatine; carnosine; carnitine
MeSH Terms: interventions — Diet, Vegetarian; Creatine; beta-Alanine

STUDY DESIGN:
Intervention Model Description: The study was scheduled over a period of 6 months. Of the 40 subjects, 10 women will continue their omnivorous diet throughout the entire study (controls) and the other 30 subjects will switch to a lacto-ovo-vegetarian diet for 6 months. The vegetarian group will be split in 2 groups, matched for age, weight, height and baseline carnosine concentrations in soleus and gastrocnemius medialis muscles. Fifteen of them will be supplemented with beta-alanine and creatine (Veg+Suppl) and the other 15 women will receive a placebo (Veg+Pla).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: A co-worker, not involved in the study design and analysis, will perform the randomisation and will prepare the containers with supplements. Only the control group will know that they are part of the control group (continuing omnivorous diet). For the vegetarian groups, subject will not know whether they are in the supplemented group or not because placebo supplements will be used
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): continued their omnivorous diet throughout the entire study
- Veg+Pla (Experimental): vegetarian + placebo: switch to a lacto-ovo-vegetarian diet for 6 months and are supplemented with placebo pills instead of beta-alanine and creatine
  Interventions: Behavioral: Vegetarian diet; Dietary Supplement: Placebo
- Veg+ creatine and beta-alanine (Experimental): switch to a lacto-ovo-vegetarian diet for 6 months and are supplemented with 1 g of creatine monohydrate (2 capsules of 500 mg) and 0.8 g of beta-alanine (1 Carnosyn® tablet) each day
  Interventions: Behavioral: Vegetarian diet; Dietary Supplement: creatine; Dietary Supplement: Beta-alanine

INTERVENTIONS:
Behavioral: Vegetarian diet
  Other Names: lacto-ovo-vegetarian diet
  Arms: Veg+ creatine and beta-alanine; Veg+Pla
Dietary Supplement: creatine — 1g creatine/day
  Arms: Veg+ creatine and beta-alanine
Dietary Supplement: Placebo — pills
  Arms: Veg+Pla
Dietary Supplement: Beta-alanine — 0.8g beta-alanine per day
  Arms: Veg+ creatine and beta-alanine

SUMMARY:
Balanced vegetarian diets are popular and contain health-promoting characteristics. A balanced lacto-ovo-vegetarian diet differs in nutrient intake from an omnivorous diet, e.g. by increased intake of fibre, magnesium and antioxidants, but lower intake of omega-3 fatty acids and vitamin B12. However, the impact of reduced to near absent intake of carnitine, carnosine and creatine in a vegetarian diet is less well established and could be relevant in relation to muscle function, exercise capacity and sports performance. Few longitudinal intervention studies investigating the effect of a vegetarian diet on the availability of these compounds currently exist.

This study aimed therefore to investigate the effect of of transiently switching omnivores onto a vegetarian diet for 6 months on muscle and plasma creatine, carnitine and carnosine homeostasis.

We hypothesized that homeostasis of creatine and carnosine would be disrupted when their dietary intake was missing. For carnitine, however, we hypothesized that homeostasis can be maintained given its slow turnover rate and its presence in some non-meat nutrients. A second aim was to investigate whether supplementation of creatine and beta-alanine (the rate-limiting precursor of carnosine synthesis), concurrently with a lacto-ovo-vegetarian diet, was able to correct for potentially emerging deficiencies.

DETAILED DESCRIPTION:
Forty healthy female omnivores will be included in this 6-month intervention study. Exclusion criteria are smoking, chronic use of medication, athletes participating in competitions, vegetarianism or eating meat or fish less than 5 times a week. The study is scheduled over a period of 6 months and measurements will be performed 1 week prior to the intervention (0M), after 3 months (3M) and within the last week (6M). Ten women will continue their omnivorous diet throughout the entire study (controls) and the other 30 subjects will switch to a lacto-ovo-vegetarian diet for 6 months. The vegetarian group will be split in 2 groups, matched for age, weight, height and baseline carnosine concentrations in soleus and gastrocnemius medialis muscles. Fifteen of them will be supplemented with beta-alanine and creatine (Veg+Suppl) and the other 15 women will receive a placebo (Veg+Pla). A co-worker, not involved in the study design and analysis, will perform the randomisation and will prepare the containers with supplements. With regard to supplementation, the study is double-blind placebo-controlled. The lacto-ovo-vegetarian diet consists of vegetables, fruits, seeds, grains, meat substitutes, eggs and dairy products and the exclusion of meat, poultry and fish. Subjects will complete a 3 day food diary at the start and after 3 months and will receive nutritional advice by a dietician during the study to prevent deficiencies in macronutrients and micronutrients. Furthermore, vegetarian recipes will be provided by email to support the subjects in their vegetarian diet.

The supplementation protocol includes simultaneously daily oral administration of creatine monohydrate (Creapure®, AlzChem AG, Germany) and slow-release beta-alanine (Carnosyn®, Natural Alternatives International, San Marcos, USA) or a placebo (maltodextrin, Natural spices, France). The supplements are considered as safe and efficacious. The Veg+Suppl group ingests 1 g of creatine monohydrate (2 capsules of 500 mg) and 0.8 g of beta-alanine (1 Carnosyn® tablet) each day during the intervention period. The Veg+Pla group will be supplemented with an identical number of capsules and tablets of maltodextrin. All subjects are asked not to take any other supplements than those provided by the current study. Compliance will be checked by asking the subjects to return the containers and counting the pills that are left. The control group, who will remain on an omnivorous diet, will not receive any supplements.

Before (0M), after 3 (3M) and 6 months (6M), subjects will perform an incremental cycling test, a fasted venous blood sample and 24hr urine will be collected, a muscle biopsy of the vastus lateralis muscle will be taken and muscle carnosine content will be determined by 1H-MRS.

A two-way analysis of variance (ANOVA) will be used to evaluate plasma and urinary metabolite concentrations, muscle carnosine, muscle biopsy metabolite concentrations, time to exhaustion (TTE) and VO2max with 'group' (Veg+Suppl; Veg+Pla; control) as between-subject factor and 'time' (0M; 3M; 6M) as within-subject factor (SPSS statistical software, SPSS Inc, Chicago, USA). For the analysis of capillary lactate and pH, measurements before and after the incremental cycling test were included as another within factor (start; end). In case of significance, analyses were repeated for each group separately and pairwise comparisons were used to compare the different time points. Values will be presented as mean ± SD and statistical significance threshold will be set at p ≤0.05.

ELIGIBILITY:
Inclusion Criteria:

* women

Exclusion Criteria:

* smoking, chronic use of medication or taking supplements, athletes participating in competitions, vegetarianism or eating meat or fish less than 5 times a week

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wim Derave, Professor, Principal Investigator — University Ghent

IPD SHARING:
Plan to Share IPD: No
individual data will not be made available to other researchers

REFERENCES:
- [Derived] Van Dyck D, Herman K, Poppe L, Crombez G, De Bourdeaudhuij I, Gheysen F. Results of MyPlan 2.0 on Physical Activity in Older Belgian Adults: Randomized Controlled Trial. J Med Internet Res. 2019 Oct 7;21(10):e13219. doi: 10.2196/13219. PMID 31593541
- [Derived] Blancquaert L, Baguet A, Bex T, Volkaert A, Everaert I, Delanghe J, Petrovic M, Vervaet C, De Henauw S, Constantin-Teodosiu D, Greenhaff P, Derave W. Changing to a vegetarian diet reduces the body creatine pool in omnivorous women, but appears not to affect carnitine and carnosine homeostasis: a randomised trial. Br J Nutr. 2018 Apr;119(7):759-770. doi: 10.1017/S000711451800017X. PMID 29569535

RESULTS

PARTICIPANT FLOW:
Groups:
- Veg+Pla: vegetarian + placebo: switch to a lacto-ovo-vegetarian diet for 6 months and are supplemented with placebo pills instead of beta-alanine and creatine
  Vegetarian diet
  Placebo: pills
- Veg+Suppl: switch to a lacto-ovo-vegetarian diet for 6 months and are supplemented with 1 g of creatine monohydrate (2 capsules of 500 mg) and 0.8 g of beta-alanine (1 Carnosyn® tablet) each day
  Vegetarian diet
  creatine and beta-alanine
Period: 0-3 Months
Arm/Group | Control | Veg+Pla | Veg+Suppl
Started | 10 | 15 | 15
Completed | 10 | 15 | 14
Not Completed | 0 | 0 | 1
Period: 3-6 Months
Arm/Group | Control | Veg+Pla | Veg+Suppl
Started | 10 | 15 | 14
Completed | 10 | 15 | 14
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Veg+Pla | Veg+Suppl | Total
Number analyzed (Participants) | 10 | 15 | 15 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.9 (9) | 26.1 (7.5) | 25.5 (6.6) | 25.6 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 15 | 15 | 40
  Male | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 10 | 15 | 15 | 40
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 10 | 15 | 15 | 40

OUTCOME MEASURES:

1. Primary Outcome: Fasted Plasma Beta-alanine Concentration
Description: Fasted venous plasma beta-alanine concentration (precursor for carnosine) at 0, 3 and 6 months of the intervention
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: µM
Arm/Group | Control | Veg+Pla | Veg+Suppl
Number analyzed (Participants) | 10 | 15 | 14
µM
  Basline | 3.37 (1.96) | 5.19 (2.26) | 4.56 (2.74)
  3 months | 3.76 (2.58) | 5.11 (1.99) | 5.8 (3.24)
  6 months | 3.9 (2.88) | 5.59 (2.63) | 5.42 (3.99)

2. Primary Outcome: Gastrocnemius Carnosine Concentration
Description: Gastrocnemius carnosine concentration at 0, 3 and 6 months of the intervention
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mM
Groups:
- Veg+ Creatine and Beta-alanine: switch to a lacto-ovo-vegetarian diet for 6 months and are supplemented with 1 g of creatine monohydrate (2 capsules of 500 mg) and 0.8 g of beta-alanine (1 Carnosyn® tablet) each day
  Vegetarian diet
  creatine: 1g creatine/day
  Beta-alanine: 0.8g beta-alanine per day
Arm/Group | Control | Veg+Pla | Veg+ Creatine and Beta-alanine
Number analyzed (Participants) | 10 | 15 | 14
mM
  Baseline | 5.18 (1.21) | 5.16 (1.46) | 5.1 (1.61)
  3 months | 5.58 (0.97) | 5.55 (1.4) | 6.55 (1.53)
  6 months | 5.68 (1.07) | 5.81 (1.82) | 7.19 (2.11)

3. Primary Outcome: Soleus Carnosine Concentration
Description: Soleus carnosine concentration at 0, 3 and 6 months of the intervention
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mM
Arm/Group | Control | Veg+Pla | Veg+Suppl
Number analyzed (Participants) | 10 | 15 | 14
mM
  Baseline | 3.91 (0.43) | 3.53 (0.94) | 3.7 (1.08)
  3 months | 3.84 (0.74) | 3.36 (0.97) | 4.72 (1.11)
  6 months | 4.0 (0.72) | 3.65 (1.38) | 4.67 (1.38)

4. Primary Outcome: Plasma Creatine Concentration
Description: Plasma creatine concentration at 0, 3 and 6 months of the intervention
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Control | Veg+Pla | Veg+Suppl
Number analyzed (Participants) | 10 | 15 | 14
µmol/L
  Baseline | 35.7 (19.8) | 29.7 (15.3) | 27.3 (9.6)
  3 months | 28.1 (11.9) | 15.8 (10.0) | 56.9 (36.3)
  6 months | 40.6 (21.6) | 16.1 (7.9) | 80.7 (65.7)

5. Primary Outcome: Plasma Creatinine Concentration
Description: Plasma creatinine at 0, 3 and 6 months of the intervention
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Control | Veg+Pla | Veg+Suppl
Number analyzed (Participants) | 10 | 15 | 14
µmol/L
  Baseline | 97.33 (7.8) | 79.49 (29.09) | 79.9 (15.83)
  3 months | 96.62 (15.1) | 85.68 (30.94) | 78.47 (17.8)
  6 months | 96.18 (17.5) | 75.41 (26.35) | 88.13 (17.09)

6. Primary Outcome: Plasma Guanidinoacetate Concentration
Description: Plasma guanidinoacetate at 0, 3 and 6 months of the intervention
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Control | Veg+Pla | Veg+Suppl
Number analyzed (Participants) | 10 | 15 | 14
µmol/L
  Baseline | 2.23 (0.49) | 2.06 (0.59) | 1.95 (0.52)
  3 months | 2.2 (0.55) | 2.05 (0.63) | 1.87 (0.72)
  6 months | 2.42 (0.92) | 2.0 (0.63) | 1.75 (0.67)

7. Primary Outcome: Urinary Creatinine Concentration
Description: Urinary creatinine at 0, 3 and 6 months of the intervention
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mg/24h
Arm/Group | Control | Veg+Pla | Veg+Suppl
Number analyzed (Participants) | 10 | 15 | 14
mg/24h
  Baseline | 1298.62 (269.46) | 1235.99 (233.05) | 1254.65 (243.38)
  3 months | 1258.78 (680.31) | 1034.3 (220.92) | 1279.41 (215.92)
  6 months | 990.25 (298.77) | 941.71 (114.46) | 1090.67 (235.57)

8. Primary Outcome: Muscle Creatine Concentration
Description: Muscle total creatine concentration in vastus lateralis muscle at 0 and 3 months of the intervention
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: mmol/kg
Arm/Group | Control | Veg+Pla | Veg+Suppl
Number analyzed (Participants) | 10 | 15 | 14
mmol/kg
  Baseline | 133.2 (11.6) | 153.5 (24.0) | 128.2 (14.9)
  3 months | 142.2 (12.7) | 128.8 (11.6) | 140.7 (17.4)

9. Primary Outcome: Plasma Carnitine Concentration
Description: plasma free carnitine concentration at 0, 3 and 6 months of the intervention
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Control | Veg+Pla | Veg+Suppl
Number analyzed (Participants) | 10 | 15 | 14
µmol/L
  Baseline | 30.81 (6.6) | 29.82 (4.45) | 28.39 (6.38)
  3 months | 28.7 (6.11) | 26.45 (6.21) | 25.71 (6.22)
  6 months | 31.71 (6.75) | 28.23 (4.88) | 27.31 (7.8)

10. Primary Outcome: Plasma Acetylcarnitine Concentration
Description: plasma acetylcarnitine concentration at 0, 3 and 6 months of the intervention
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Control | Veg+Pla | Veg+Suppl
Number analyzed (Participants) | 10 | 15 | 14
µmol/L
  Baseline | 8.49 (2.24) | 7.71 (1.95) | 8.09 (1.98)
  3 months | 6.82 (1.31) | 6.93 (1.78) | 6.77 (1.33)
  6 months | 7.15 (1.41) | 7.54 (1.67) | 7.15 (3.16)

11. Primary Outcome: Plasma Total Carnitine Concentration
Description: plasma total carnitine concentration (free + acetyl) at 0, 3 and 6 months of the intervention
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Control | Veg+Pla | Veg+Suppl
Number analyzed (Participants) | 10 | 15 | 14
µmol/L
  Baseline | 41.58 (6.97) | 40.85 (7.42) | 40.24 (5.75)
  3 months | 37.96 (6.44) | 36.16 (7.83) | 35.9 (5.48)
  6 months | 41.25 (8.02) | 38.58 (6.45) | 37.87 (9.51)

12. Primary Outcome: Muscle Carnitine Concentration
Description: muscle free carnitine concentration in vastus lateralis muscle at 0 and 3 months of the intervention
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: mmol/kg dry weight
Arm/Group | Control | Veg+Pla | Veg+Suppl
Number analyzed (Participants) | 10 | 15 | 14
mmol/kg dry weight
  Baseline | 13.1 (4.0) | 12.1 (4.1) | 10.7 (2.8)
  3 months | 11.5 (2.9) | 11.5 (4.9) | 9.7 (3.2)

13. Primary Outcome: Muscle Acetylcarnitine Concentration
Description: muscle acetylcarnitine concentration in vastus lateralis muscle at 0 and 3 months of the intervention
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: mmol/kg dry weight
Arm/Group | Control | Veg+Pla | Veg+Suppl
Number analyzed (Participants) | 10 | 15 | 14
mmol/kg dry weight
  Baseline | 3.3 (3.2) | 4.2 (2.4) | 3.3 (2.9)
  3 months | 3.6 (1.9) | 3.5 (4.1) | 3.2 (2.5)

14. Primary Outcome: Muscle Total Carnitine Concentration
Description: muscle total carnitine concentration (free + acetylcarnitine) in vastus lateralis muscle at 0 and 3 months of the intervention
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: mmol/kg dry weight
Arm/Group | Control | Veg+Pla | Veg+Suppl
Number analyzed (Participants) | 10 | 15 | 14
mmol/kg dry weight
  Baseline | 16.5 (2.4) | 16.3 (3.5) | 13.9 (2.3)
  3 months | 15.5 (3.2) | 13.6 (2.3) | 12.7 (2.2)

15. Secondary Outcome: Vitamin D Status
Description: Serum 25-Hydroxyvitamin D concentration at 0, 3 and 6 months of the intervention
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Control | Veg+Pla | Veg+Suppl
Number analyzed (Participants) | 10 | 15 | 14
ng/ml
  Baseline | 32.7 (13.6) | 29.1 (10.3) | 29.8 (8.9)
  3 months | 24.9 (10.0) | 22.7 (9.0) | 24.6 (7.8)
  6 months | 34.6 (14.1) | 30.1 (10.8) | 31.1 (9.1)

16. Secondary Outcome: Urinary Biomarker for Meat Intake: Pi-methyl-histidine
Description: urinary pi-methyl-histidine concentration at 0, 3 and 6 months of the intervention
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mg/24h
Arm/Group | Control | Veg+Pla | Veg+Suppl
Number analyzed (Participants) | 10 | 15 | 14
mg/24h
  Baseline | 161.9 (111.2) | 167.4 (145.3) | 212.9 (201.0)
  3 months | 117.8 (124.8) | 26.4 (10.7) | 28.7 (9.1)
  6 months | 122.5 (168.8) | 15.1 (4.7) | 18.0 (6.7)

17. Secondary Outcome: Urinary Biomarker for Meat Intake: Tau-methyl-histidine
Description: urinary tau-methyl-histidine concentration at 0, 3 and 6 months of the intervention
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mg/24h
Arm/Group | Control | Veg+Pla | Veg+Suppl
Number analyzed (Participants) | 10 | 15 | 14
mg/24h
  Baseline | 55.2 (25.3) | 63.1 (20.0) | 63.0 (22.3)
  3 months | 74.6 (61.6) | 43.1 (15.3) | 46.1 (16.0)
  6 months | 42.6 (21.5) | 27.6 (7.1) | 26.5 (8.5)

18. Secondary Outcome: Urinary Biomarker for Meat Intake: Anserine
Description: urinary anserine concentration at 0, 3 and 6 months of the intervention
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mg/24h
Arm/Group | Control | Veg+Pla | Veg+Suppl
Number analyzed (Participants) | 10 | 15 | 14
mg/24h
  Baseline | 15.0 (14.3) | 9.2 (7.9) | 10.7 (12.9)
  3 months | 9.5 (7.4) | 5.5 (2.9) | 4.4 (2.2)
  6 months | 11.6 (23.2) | 4.0 (1.9) | 2.6 (1.1)

19. Secondary Outcome: VO2max
Description: VO2max during incremental cycling test performed at 0, 3 and 6 months
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: ml/min/kg
Arm/Group | Control | Veg+Pla | Veg+Suppl
Number analyzed (Participants) | 10 | 15 | 14
ml/min/kg
  Baseline | 40.4 (6.4) | 39.4 (6.4) | 36.6 (6.3)
  3 months | 39.0 (8.8) | 37.8 (8.0) | 34.8 (4.7)
  6 months | 39.4 (6.9) | 38.1 (6.6) | 34.5 (4.9)

20. Secondary Outcome: Time to Exhaustion
Description: Time to exhaustion during incremental cycling test performed at 0, 3 and 6 months
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Control | Veg+Pla | Veg+Suppl
Number analyzed (Participants) | 10 | 15 | 14
minutes
  Baseline | 14.5 (1.9) | 15.1 (2.7) | 13.8 (2.6)
  3 months | 14.0 (3.0) | 14.7 (2.5) | 13.6 (2.4)
  6 months | 14.6 (2.2) | 15.0 (2.5) | 13.8 (2.9)

21. Secondary Outcome: Capillary Lactate
Description: capillary lactate at the start and at the end of the incremental cycling test performed at 0, 3 and 6 months
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Control | Veg+Pla | Veg+Suppl
Number analyzed (Participants) | 10 | 15 | 14
mmol/L
  Baseline - start | 1.9 (0.5) | 2.0 (0.7) | 1.8 (0.8)
  Baseline - end | 10.7 (1.6) | 12.4 (4.2) | 10.7 (2.7)
  3 months - start | 2.4 (1.0) | 2.0 (0.9) | 2.2 (0.9)
  3 months - end | 11.4 (2.6) | 14.1 (2.1) | 12.2 (2.3)
  6 months - start | 2.0 (0.5) | 1.7 (0.4) | 2.2 (1.1)
  6 months - end | 12.1 (2.0) | 12.7 (1.1) | 13.1 (2.1)

22. Secondary Outcome: Capillary pH
Description: capillary pH at the start and at the end of the incremental cycling test performed at 0, 3 and 6 months
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Control | Veg+Pla | Veg+Suppl
Number analyzed (Participants) | 10 | 15 | 14
pH
  Baseline - start | 7.4 (0.02) | 7.41 (0.02) | 7.42 (0.02)
  Baseline - end | 7.28 (0.03) | 7.24 (0.07) | 7.28 (0.06)
  3 months - start | 7.4 (0.03) | 7.42 (0.03) | 7.41 (0.01)
  3 months - end | 7.27 (0.04) | 7.23 (0.04) | 7.26 (0.04)
  6 months - start | 7.42 (0.04) | 7.43 (0.02) | 7.43 (0.01)
  6 months - end | 7.29 (0.05) | 7.27 (0.03) | 7.28 (0.04)

ADVERSE EVENTS:
Arm/Group | Control | Veg+Pla | Veg+Suppl
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/15 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/15 | 0/14
Other Adverse Events (participants affected / at risk) | 0/10 | 0/15 | 0/14

LIMITATIONS AND CAVEATS:
A far too low number of subjects consented to have muscle biopsies taken at 6M. Therefore, muscle analyses were restricted to the 0 and 3M time points.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes